CLINICAL TRIAL: NCT00093873
Title: A Phase 1, First in Human, Open-Label, Dose Finding Study Evaluating the Safety and Pharmacokinetics of AMG 706 in Subjects With Advanced Solid Tumors
Brief Title: Study Evaluating AMG 706 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030116
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Tumors
Keywords: Cancer; antiangiogenesis; Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Angiogenesis Inhibitors; motesanib diphosphate

ARMS (1):
- AMG 706 (Experimental): AMG 706 QD
  Interventions: Drug: Anti-angiogenesis; Drug: AMG 706

INTERVENTIONS:
Drug: Anti-angiogenesis — Anti-angiogenesis
Drug: AMG 706 — Anti-angiogenesis

SUMMARY:
This study will determine the safety and pharmacokinetics of AMG 706 in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria: Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2003-07; Primary Completion 2006-02 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | Cycle 1

SECONDARY OUTCOMES:
Dose selection | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Rosen LS, Kurzrock R, Mulay M, Van Vugt A, Purdom M, Ng C, Silverman J, Koutsoukos A, Sun YN, Bass MB, Xu RY, Polverino A, Wiezorek JS, Chang DD, Benjamin R, Herbst RS. Safety, pharmacokinetics, and efficacy of AMG 706, an oral multikinase inhibitor, in patients with advanced solid tumors. J Clin Oncol. 2007 Jun 10;25(17):2369-76. doi: 10.1200/JCO.2006.07.8170. PMID 17557949
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_63_AMG_706_20030116.pdf